CLINICAL TRIAL: NCT03549377
Title: Neural Correlates of the Associations Between Sleep Functioning, Self-regulation, Academic Functioning, and Problem Behaviors
Brief Title: Neural Correlates of Self-regulation on Academic Functioning
Status: Completed | Type: Observational
Sponsor: Alexander Vazsonyi (Other)
Responsible Party: Sponsor-Investigator, Alexander Vazsonyi, Endowed Professor, University of Kentucky
Organization: University of Kentucky (Other)
Other Study IDs: 44065
Record Dates: First submitted 2018-05-14; First posted 2018-06-08 (Actual); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: Self-Control
Keywords: Sleep; Academic functioning; Problem behaviors; College age youth; Self-regulation
MeSH Terms: conditions — Self-Control; Problem Behavior

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Rested: Based on Pittsburgh Sleep Quality Index, participants scoring in the top 10-20% will be assigned to the rested group and will experience deception as part of the delayed gratification task
  Interventions: Behavioral: Deception
- Sleep-deprived: Based on Pittsburgh Sleep Quality Index, participants scoring in the bottom 10-20% will be assigned to the sleep-deprived group and will experience deception as part of the delayed gratification task
  Interventions: Behavioral: Deception

INTERVENTIONS:
Behavioral: Deception — Participants will be deceived during delayed gratification task.

SUMMARY:
The main objectives of the study include: 1. What are the differences in self-regulation and its neurophysiological and neuroanatomical correlates between college students with poor and excellent sleep functioning? 2. Does sleep functioning (assessed both by questionnaires and actigraphy), and self-control/self-regulation (questionnaire and imaging data) predict academic achievement and problem behaviors in college students?

DETAILED DESCRIPTION:
Based on the Self-Control Theory, individual differences in characteristics such as impulsivity, risk-seeking, and self-regulation consistently predict health-compromising and problem behaviors as well as academic functioning and success in adolescents and young adults.[1] Although suboptimal self-regulation is normative in adolescence and young adulthood, [2] it might result in negative consequences for adolescents' and young adults' health and well-being, including substance use, school/college dropout, or troubles with law. A recent line of research suggested that self-regulation problems are associated with insufficient and poor sleep.[3] As adolescents and young adults frequently report poor sleep functioning,[4] their self-regulation abilities might be further compromised by unfavorable sleep functioning with consequences for youths' problem behaviors and academic success. To mitigate this problem, some efforts have followed to ensure that adolescents get enough quality sleep (e.g., delayed school start times). However, the associations between sleep functioning, self-regulation, academic functioning, and problem behaviors were established predominantly using questionnaire data. Neurophysiological correlates of these associations have not been extensively studied. In the proposed study, this gap in scholarship will be addressed by linking sleep functioning to self-regulation indicated by neuropsychological and neuroanatomical data, and predicting academic achievement and problem behaviors with sleep and self-regulation. This explorative, pilot study is a first step in efforts to understand the issue; it will be carried out with a college student sample (N = 48, 50% female) which will also have implications for future research focused on adolescents (middle and high school students). Pilot data will inform the development of a larger study that will include adolescents (middle and high school students) and will support grant applications. Results will have a potential for prevention /intervention programs and policy targeting youth, such as school start times setting. This study will be carried out as a collaboration between the Department of Family Sciences at the University of Kentucky and the Department of Human Development and Family Studies at the Texas Tech University. Data will be collected following the same procedures described in this application both at the University of Kentucky and Texas Tech campuses. Research team at the Texas Tech University has submitted their own Institutional Review Board (IRB) application that is now being reviewed.

ELIGIBILITY:
Inclusion Criteria:

Healthy college-age youth between the ages of 18 and 24 years

Exclusion Criteria:

* Gross impairment of vision or hearing
* Inability to read and follow written instructions
* Physical, neurological, or concurrent psychiatric impairments
* Regular intake of psychotropic medication (such as methylphenidate used to treat Attention Deficit Hyperactivity Disorder (ADHD), antidepressants, or anti-anxiety medication)
* A history of head injury that resulted in loss of consciousness/a history of brain surgery/or seizures
* A current/past history of smoking and/or alcohol or drug abuse (i.e., five or more drinks in one sitting or 15 drinks or more during a week for men, and four drinks on one occasion or eight drinks over the course of a week for women; additionally, regular drug use, including marijuana)
* Current pregnancy
* Any metallic objects in your body (such as braces, pacemakers, surgical devices, piercings that cannot be removed etc.) Enrollment of the subjects will start in May 2018 and will be finished by the end of December 2018.

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study sample will consist of 24 healthy college students (12 males and 12 females) between ages 18 - 24 years.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2018-05-11 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
Rested versus sleep deprived group differences of Functional magnetic resonance imaging (fMRI) Blood oxygenation level dependent (BOLD) responses for Stop Signal Reaction Time Task (SSRT) Stop Signals | Up to 45 days following selection for inclusion based on prescreen, cross-sectional study
  Rested versus sleep deprived group differences of functional magnetic resonance imaging reactivity of the whole brain while performing a Stop Signal Reaction Time Task
Rested versus sleep deprived group differences of fMRI BOLD responses for a Go-NoGo Continuous Performance Task (CPT) | Up to 45 days following selection for inclusion based on prescreen, cross-sectional study
  Rested versus sleep deprived group differences of functional magnetic resonance imaging reactivity of the whole brain while performing a Go-NoGo Continuous Performance Task
Rested versus sleep deprived group differences of brain structural connectivity | Up to 45 days following selection for inclusion based on prescreen, cross-sectional study
  Rested versus sleep deprived group differences of brain structural connectivity as measured by diffusion tensor imaging and analyzed using tract-based spatial statistics
Rested versus sleep deprived group differences of brain structure | Up to 45 days following selection for inclusion based on prescreen, cross-sectional study
  Rested versus sleep deprived group differences of brain structure as determined by voxel based morphometry of structural magnetic resonance imaging data

OTHER OUTCOMES:
Rested versus sleep deprived group differences in sleep time preferences | Up to 45 days following selection for inclusion based on prescreen, cross-sectional study
  Morningness-eveningness Questionnaire
Rested versus sleep deprived group differences in hours of sleep | Up to 45 days following selection for inclusion based on prescreen, cross-sectional studyUp to 45 days following selection for inclusion based on prescreen, cross-sectional study
  Sleep quantity
Rested versus sleep deprived group differences in low self-control | Up to 45 days following selection for inclusion based on prescreen, cross-sectional study
  Low Self-Control Scale (LSC)
  * Low self-control scale (24 items) measures low self-control.
  * The total score ranges from 1 to 5.
  * Five subscales called impulsivity, simple tasks, risk seeking, physical activities, self-centered, and temper, each provide subscale score ranging from 1 to 5.
  * Higher values indicate higher lower self-control, in other words, worse outcomes.
  * A total score is developed by averaging all 24 items across all subscales. Subscale scores also represent the averaged responses to their corresponding items.
Rested versus sleep deprived group differences in sensation seeking and impulsivity | Up to 45 days following selection for inclusion based on prescreen, cross-sectional study
  Zuckerman Impulsivity and Sensation Seeking Scale
  * Impulsivity and Sensation Seeking Scale (19 items) measures impulsivity and sensation seeking.
  * Total score ranges from 0 to 19. Impulsivity (i.e., one of the two subscales) score ranges from 0 to 8 (8 items), whereas Sensation Seeking score ranges from 0 to 11 (11 items).
  * For total as well as for each subscale scores, higher values indicate more impulsivity and sensation seeking, respectively.
  * Total and subscale scores are computed by summing the responses (19, 11, and 8 items respectively).
Rested versus sleep deprived group differences in internalizing behaviors | Up to 45 days following selection for inclusion based on prescreen, cross-sectional study
  Weinberger Adjustment Inventory
Rested versus sleep deprived group differences in deviance/externalizing subscales | Up to 45 days following selection for inclusion based on prescreen, cross-sectional study
  Normative Deviance Scale, Short Form
  * Normative Deviance Scale-Short Form (21 items); the scale measures involvement in deviant and norm-violating behaviors.
  * Total scores range from 1 to 5. Seven subscale scores (i.e., vandalism, alcohol use, drug use, school misconduct, general deviance, theft, assault) each range from 1 to 5, 3 items each.
  * Higher scores indicate greater deviance (more frequent involvement), in other word, worse outcome.
  * A total score, as well as subscale scores, are computed by averaging responses of the corresponding items.
Rested versus sleep deprived group differences in GPA/SAT/ACT Scores | Up to 45 days following selection for inclusion based on prescreen, cross-sectional study
  Grade point average (GPA)/Scholastic Aptitude Test (SAT)/American College Test (ACT) Score
Academic Dishonesty Scale | Up to 45 days following selection for inclusion based on prescreen, cross-sectional study
  Rested versus sleep deprived group differences in school attitudes
Rested versus sleep deprived group differences in academic concentration | Up to 45 days following selection for inclusion based on prescreen, cross-sectional study
  Academic Concentration Measure
Rested versus sleep deprived group differences in academic aspirations and expectations | Up to 45 days following selection for inclusion based on prescreen, cross-sectional study
  Academic Expectations and Aspirations
Rested versus sleep deprived group differences in school attitudes | Up to 45 days following selection for inclusion based on prescreen, cross-sectional study
  School Attitudes Assessment Survey
Rested versus sleep deprived group differences in Flanker Inhibitory Control and Attention Test, Dimensional Change Card Sort Test, List Sorting Working Memory Test | Up to 45 days following selection for inclusion based on prescreen, cross-sectional study
  NIH toolbox Cognition Battery
Rested versus sleep deprived group differences in Flanker Inhibitory Control and Attention Test, Dimensional Change Card Sort Test, Picture Sequence Memory Test, | Up to 30 days following selection for inclusion based on prescreen, cross-sectional study
  NIH toolbox Cognition Battery
Rested versus sleep deprived group differences in commission errors in Balloon Analogue Risk Task (BART), , omission errors | Up to 30 days following selection for inclusion based on prescreen, cross-sectional study
  Balloon Analogue Risk Task (BART)
Rested versus sleep deprived group differences in commission errors in a Go-NoGo CPT, omission errors | Up to 30 days following selection for inclusion based on prescreen, cross-sectional study
  Go/NoGo continuous performance task (CPT)

CONTACTS AND LOCATIONS:
Overall Officials: Alexander T Vazsonyi, Ph.D., Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No
No plan at this time

REFERENCES:
- [Background] Gottfredson MR, Hirschi T. A general theory of crime. Stanford: Stanford University Press; 1990.
- [Background] Steinberg L, Albert D, Cauffman E, Banich M, Graham S, Woolard J. Age differences in sensation seeking and impulsivity as indexed by behavior and self-report: evidence for a dual systems model. Dev Psychol. 2008 Nov;44(6):1764-78. doi: 10.1037/a0012955. PMID 18999337
- [Background] Owens JA, Dearth-Wesley T, Lewin D, Gioia G, Whitaker RC. Self-Regulation and Sleep Duration, Sleepiness, and Chronotype in Adolescents. Pediatrics. 2016 Dec;138(6):e20161406. doi: 10.1542/peds.2016-1406. Epub 2016 Nov 3. PMID 27940688
- [Background] Wheaton AG, Jones SE, Cooper AC, Croft JB. Short Sleep Duration Among Middle School and High School Students - United States, 2015. MMWR Morb Mortal Wkly Rep. 2018 Jan 26;67(3):85-90. doi: 10.15585/mmwr.mm6703a1. PMID 29370154